CLINICAL TRIAL: NCT00468663
Title: Ambient Air Pollution, Preeclampsia, and Preterm Delivery
Status: Completed | Type: Observational
Sponsor: National Institute of Environmental Health Sciences (NIEHS) (NIH)
Other Study IDs: 14716-CP-001
Record Dates: First submitted 2007-05-02; First posted 2007-05-03 (Estimated); Last update posted 2015-04-14 (Estimated); Status verified 2015-04

CONDITIONS: Preeclampsia; Preterm Delivery
Keywords: preeclampsia; preterm delivery; lipid peroxidation; inflammation
MeSH Terms: conditions — Pre-Eclampsia; Premature Birth; Inflammation

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
An epidemiologic study of pregnant women in western Washington to measure the relationships between exposure to air pollutants and risks of preeclampsia and preterm delivery.

DETAILED DESCRIPTION:
We will design models that use local traffic, weather, and population characteristics to predict monthly ambient concentrations of fine particulate matter (PM2.5) and carbon monoxide (CO). These models will be used to estimate study participants' PM2.5 and CO exposures during and before pregnancy. We will test whether these air pollutant exposures are associated with subsequent risk of preeclampsia and preterm delivery. Additionally, we will test biological markers of maternal lipid peroxidation (thiobarbituric acid reactive substances) and inflammation (high sensitivity C-reactive protein) in maternal blood samples drawn during early pregnancy. We will also examine carboxyhemoglobin measured in early-pregnancy maternal blood samples as a marker of CO exposure.

ELIGIBILITY:
Inclusion Criteria:

* English speaking
* enrolled in parent study
* pregnant at <20 weeks gestation and attending prenatal care clinics affiliated with Swedish Medical Center and Tacoma General Hospital

Exclusion Criteria:

-

Min Age: 18 Years
Age Groups: Adult, Older Adult
Enrollment: 4200 (Actual)
Dates: Start 2006-07; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carole Rudra, Ph.D, MPH, Principal Investigator — Swedish Medical Center, First Hill; Michelle A Williams, Sc.D, Principal Investigator — Swedish Medical Center